Date: April 9, 2019

Title: Importance of sock type in the development of foot lesions on low-difficulty, short hikes.

**Description of document:** The document describe, among other things, the purpose, the procedures, the risks and the potential benefits of study. It was approved by the committee etica of University Extremadura like part a project general entitled "Ruta de la Plata por Cáceres. A healthy way".

| INFORMATION | TO THE | PATIFNT | AND INFOR | MED CONSENT |
|-------------|--------|----------|-----------|---------------|
| | 10 111 | INITIALI | AND INTOK | MILD COMPLIAT |

| Date: | Name and surnar | ne | DNI | Number of ( | dorsal |
|-------|-----------------|----|-----|-------------|--------|

You have been invited to participate in a research project on the podiatric health of the hiker who walk along the route of La Plata through Cáceres. This project will focus on analyzing foot injuries that appear to the hiker during the Galisteo-Cáparra stage.

- I ACCEPT TO COLLABORATE in this investigation. If you agree to collaborate, you will be asked to participate by signing this document that will act as informed consent. You also have to fill out a survey. If you agree to participate, you must wear a training boots with specific features that we will tell you and you should know that the researchers will provide the socks that must be worn along the hike. At the beginning of the hike, you will be explored and after analyzing your podiatry characteristics, you will be provided with several hiking socks in order to study some characteristics of them as external factors damaging agents or injury protectors on your feet and start your route. Half way through, you will be explore again by the same podiatrist and treat your feet again if necessary, and at the end of the hike you will be explored again. After that, podiatric advice will be recommended if you need them. Your participation will be free and will not entail any cost to you. Participating in the study does not entail any additional risk to those inherent in the performance of a short walk and low difficulty.

The benefit you can obtain will be an individualized podiatric treatment that will guide you in the recommended preventive measures for the hiking activity proposed, in addition to its contribution indirectly, to a greater knowledge of external or internal factors that may influence pathologies that the hiker suffers when making a hike of little difficulty and short term. These results will help us to perform preventive podiatry measures for hikers.

All the data offered for this work will only be used for teaching and research purposes and will be kept anonymous to guarantee your confidentiality, right to privacy and your own image. If you have any questions or would like more information about this research, please contact Ana M<sup>a</sup> Pérez Pico, Professor at the University Center of Plasencia. UEX.

Your signature on this document means that you have decided to participate after having read and discussed the information presented on this consent form.

Name of the participant, Signature/ Date

Name of the responsible of research, Signature/Date